CLINICAL TRIAL: NCT01625039
Title: The Impact of an Employee Wellness Programme in Clothing/Textile Manufacturing Companies: A Randomised Control Trial
Brief Title: Impact of Employee Wellness Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Naila Edries, Clinical Educator, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2012-06-12; First posted 2012-06-21 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Obesity
Keywords: Occupational health; cognitive behavioural therapy; physiotherapy; physical activity
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participated in weekly educational workshops
  Interventions: Behavioral: Employee wellness programme
- Control group (Active Comparator): Received once off educational session and materials
  Interventions: Behavioral: Comparator (Once off educational session and educational materials)

INTERVENTIONS:
Behavioral: Employee wellness programme — The experimental group was subjected to a wellness programme based on the principles of cognitive behaviour therapy (CBT) as well as weekly supervised exercise classes over six weeks.
  Other Names: Exercise classes
  Arms: Intervention
Behavioral: Comparator (Once off educational session and educational materials) — Once off educational session and educational materials
  Other Names: Health education
  Arms: Control group

SUMMARY:
The introduction of a wellness programme for workers employed in a clothing factory will improve quality of life, pain, attendance at work and levels of physical activity.

DETAILED DESCRIPTION:
Introduction: The prevalence of health risk behaviours is growing amongst South African employees. Health risk behaviours have been identified as a major contributor to reduced health related quality of life (HRQoL) and the increase prevalence of non-communicable diseases. Worksite wellness programmes promise to promote behaviour changes amongst employees and to improve their HRQoL.

Aims: The aim of this study was to evaluate the short-term efficacy of an employee wellness programme on HRQoL, health behaviour change, levels of self efficacy, pain intensity, body mass index (BMI) and absenteeism amongst clothing and textile manufacturing employees.

Methods: The study was a randomised control trial consisting of 80 participants from three clothing manufacturing companies in South Africa. The experimental group was subjected to a wellness programme based on the principles of cognitive behaviour therapy (CBT) as well as weekly supervised exercise classes over six weeks. The control group received a once-off health promotion talk and various educational pamphlets, with no further intervention. Measurements were recorded at baseline and at six weeks post-intervention. Outcome measures used included the EQ-5D, Brief Pain Inventory-SF, Stanford Exercise Behaviours Scale, Stanford Self-Efficacy Scale, Stanford Self-Rated Health Scale, BMI and absenteeism.

Data Analysis: All the data were analysed with the Statistica-8 software program. Although t-tests are the most commonly used statistical method for evaluating the differences in the means between two groups (e.g. control and experimental), it assumes that the variable is normally distributed. Thus, because the ordinal data were not normally distributed, non-parametric tests were used to evaluate the differences in the medians between the two groups and to determine the level of significance. The Sign test was used in place of the paired t-test to determine the within group changes. The Mann-Whitney U test was used in place of the independent t-test to determine the difference between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* All factory workers who volunteered to take part in the study

Exclusion Criteria:

* Subjects were excluded from the study if they reported uncontrolled diabetes and hypertension, coronary heart disease or any other illness that rendered participation in the exercise component unsafe.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
EQ-5D | Baseline, change in EQ-5D at 6 weeks
  Generic Health Related Quality of Life measure

SECONDARY OUTCOMES:
Stanford Exercise Behaviour Scale | Baseline, change in stanford exercise behaviour at 6 weeks
  Self reported participation in different forms of physical exercise
Body Mass Index | Baseline, Change in BMI at 6 weeks
  Measurement of height and weight using standardized scales.
Absenteeism from work | All absenteeism during the six weeks prior, during the six weeks of intervention and six weeks post intervention
  Scrutiny of attendance records

CONTACTS AND LOCATIONS:
Overall Officials: Naila Edries, BSc, Principal Investigator — University of Cape Town
Locations (1):
- Clothing Factories, Cape Town, Observatory, South Africa

REFERENCES:
- [Derived] Edries N, Jelsma J, Maart S. The impact of an employee wellness programme in clothing/textile manufacturing companies: a randomised controlled trial. BMC Public Health. 2013 Jan 11;13:25. doi: 10.1186/1471-2458-13-25. PMID 23311458